CLINICAL TRIAL: NCT01437423
Title: Regulatory Post-Marketing Surveillance (PMS) Study for TETRAXIM™(Combined Vaccine of Adsorbed Diphtheria, Tetanus, Acellular Pertussis and Enhanced Inactivated Poliomyelitis)
Brief Title: Regulatory Post-Marketing Surveillance Study for TETRAXIM™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: E2I59; U1111-1114-7745 (Other: WHO)
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Diphtheria; Tetanus; Pertussis; Poliomyelitis
Keywords: Diphtheria; Tetanus; Pertussis; Poliomyelitis; TETRAXIM™
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis | interventions — Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TETRAXIM™ vaccine (Experimental): Participants will receive a primary or booster dose of TETRAXIM™
  Interventions: Biological: TETRAXIM™: Combined adsorbed diphtheria, tetanus, acellular pertussis and enhanced inactivated polio

INTERVENTIONS:
Biological: TETRAXIM™: Combined adsorbed diphtheria, tetanus, acellular pertussis and enhanced inactivated polio — 0.5 mL, Intramuscular at 2, 4, 6 months (Primary) or at 4 to 6 years (Booster) vaccination
  Other Names: TETRAXIM™

SUMMARY:
The purpose of this study is to assess the safety of TETRAXIM™ administered in routine clinical practice according to Korea Food and Drug Administration Notification No. 2009-46 "Basic standard for reexamination of new drug" based on the pharmaceutical law in Korea.

DETAILED DESCRIPTION:
Primary vaccination will be administered from 2 months and booster vaccination from age 4 to 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 2 months or more of age (as indicated in the currently approved local product labeling) and who are given the study vaccine at least one dose or more, during a routine health-care visit, as primary immunization or booster immunization for the prevention of diphtheria, tetanus, pertussis, poliomyelitis.
* Written informed consent obtained from the subject's parents/legal representative.

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2011-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Choe YJ, Vidor E, Manson C. Post-Marketing Surveillance of Tetravalent Diphtheria-Tetanus-Acellular Pertussis and Inactivated Poliovirus (DTaP-IPV) Vaccine in South Korea, 2009 to 2015. Infect Dis Ther. 2022 Aug;11(4):1479-1492. doi: 10.1007/s40121-022-00650-8. Epub 2022 May 14. PMID 35575974
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled for a 6 year surveillance period (31 August 2009 to 30 August 2015) at 8 clinic centers in Korea.
Pre-assignment Details: Of the 662 participants whose case report forms were retrieved, 647 participants were included in the safety analysis.
Groups:
- TETRAXIM™ Vaccination and Booster Group: Children under 12 years old who received the 3-dose primary series injection of TETRAXIM™ vaccination and booster, were enrolled during the 6-year surveillance period, and whose case report forms were retrieved.
Period: Overall Study
Arm/Group | TETRAXIM™ Vaccination and Booster Group
Started | 662
Completed | 647
Not Completed | 15
Not completed — Lost to Follow-up | 12
Not completed — Off label usage | 3

BASELINE CHARACTERISTICS:
Arm/Group | TETRAXIM™ Vaccination and Booster Group
Number analyzed (Participants) | 647
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 647
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 8.16 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 327
  Male | 320
Region of Enrollment [Number; unit: Participants]
  Korea, Republic of | 647

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Unexpected Adverse Events Up 30 Days Following A Primary Series and Booster Injection of TETRAXIM™.
Description: The number of participants reporting unexpected adverse events within 30 days following a primary series and booster injection of TETRAXIM™ (Combined vaccine of adsorbed diphtheria, tetanus, acellular pertussis and enhanced inactivated poliomyelitis)) during 6 year surveillance period.
Time Frame: Up to 30 days post-primary and booster vaccination
Population: Adverse events were reported from the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | TETRAXIM™ Vaccination and Booster Group
Number analyzed (Participants) | 647
Participants
  Bronchitis | 76
  Upper respiratory tract infection | 30
  Coryza | 10
  Bronchiolitis | 6
  Coughing | 4
  Rhinitis | 4
  Common cold | 3
  Tonsillitis | 3
  Allergic rhinitis | 1
  Asthma | 1
  Croup | 1
  Nasopharyngitis | 1
  Enteritis | 20
  Gastroenteritis | 5
  Constipation | 2
  Gastritis acute | 2
  Dermatitis contact | 15
  Dermatitis atopic | 4
  Dermatitis diaper | 3
  Rash impetiginous | 3
  Contact eczema | 1
  Dermatitis seborrhoeic | 1
  Eczema allergic | 1
  Otitis media | 5
  Hand foot and mouth disease | 1
  Conjunctivitis | 2
  Red eye | 1

2. Other Pre Specified Outcome: Number of Participants Reporting Solicited Adverse Events Following A Primary Series Injection of TETRAXIM™.
Description: Injection-site reactions: Tenderness, Erythema, and Swelling. Systemic reactions: Fever (Temperature) and Crying abnormal. Grade 3 Injection-site reactions: Tenderness, Cries when injected limb is moved or the movement of the injected limb is reduced; Erythema and Swelling, ≥5 cm. Grade 3 Systemic reactions: Fever, >39.5˚C; Crying abnormal, >3 hours.
Time Frame: Up to 30 days post-primary and booster vaccination
Population: Solicited adverse events were reported from the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | TETRAXIM™ Vaccination and Booster Group
Number analyzed (Participants) | 647
Participants
  Any Injection-site Tenderness | 20
  Grade 3 Injection-site Tenderness | 0
  Any Injection-site Erythema | 10
  Grade 3 Injection-site Erythema | 0
  Any Injection-site Swelling | 10
  Grade 3 Injection-site Swelling | 0
  Any Fever | 6
  Grade 3 Fever | 0
  Any Crying abnormal | 1
  Grade 3 Crying abnormal | 0

3. Other Pre Specified Outcome: Number of Participants Reporting Unsolicited Adverse Events Following A Primary Series and Booster Injection of TETRAXIM™.
Description: The number of participants reporting unsolicited adverse events within 30 days following a primary series and booster injection of TETRAXIM™ (Combined vaccine of adsorbed diphtheria, tetanus, acellular pertussis and enhanced inactivated poliomyelitis) during the 6 year surveillance period
Time Frame: Up to 30 days post-primary and booster of TETRAXIM™ vaccination
Population: Unsolicited adverse events were reported from the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | TETRAXIM™ Vaccination and Booster Group
Number analyzed (Participants) | 647
Participants
  Bronchitis | 79
  Upper respiratory tract infection | 32
  Coryza | 10
  Bronchiolitis | 6
  Coughing | 4
  Rhinitis | 4
  Common cold | 3
  Tonsillitis | 3
  Allergic rhinitis | 1
  Asthma | 1
  Croup | 1
  Nasopharyngitis | 1
  Enteritis | 20
  Gastroenteritis | 5
  Diarrhoea | 4
  Constipation | 2
  Gastritis acute | 2
  Vomiting | 1
  Dermatitis contact | 15
  Dermatitis atopic | 4
  Dermatitis diaper | 3
  Rash impetiginous | 3
  Contact eczema | 1
  Dermatitis seborrhoeic | 1
  Eczema allergic | 1
  Fever | 3
  Otitis media | 6
  Hand foot and mouth disease | 1
  Conjunctivitis | 2
  Red eye | 1
  Irritability | 1

4. Other Pre Specified Outcome: Occurrence of Adverse Events by Demographic Characteristic of Participants Following A Single Dose of TETRAXIM™.
Description: The number of participants reporting adverse events by demographic characteristic following a primary series injection of TETRAXIM™ (Combined vaccine of adsorbed diphtheria, tetanus, acellular pertussis and enhanced inactivated poliomyelitis) during the 6 years surveillance period is reported.
Time Frame: Up to 30 days post-primary and booster of vaccination
Population: Adverse events were reported from the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | TETRAXIM™ Vaccination and Booster Group
Number analyzed (Participants) | 647
Participants
  Gender; Male (N=320) | 82
  Gender; Female (N=327) | 99
  Age; <12 months (N=602) | 167
  Age; 48 to <60 months (N=35) | 12
  Age; 60 to <72 months (N=7) | 1
  Age; ≥72 months (N=3) | 1

ADVERSE EVENTS:
Time Frame: Adverse event data (solicited and unsolicited) were collected up to 30 days after the primary series injection of TETRAXIM™ during the 6 year surveillance period.
Arm/Group | TETRAXIM™ Vaccination and Booster Group
Serious Adverse Events (participants affected / at risk) | 0/647
Other Adverse Events (participants affected / at risk) | 79/647
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TETRAXIM™ Vaccination and Booster Group (N=647)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 79 (79)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 32 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications